CLINICAL TRIAL: NCT03557879
Title: Exome Analysis on Hearing Impaired Patients
Brief Title: Exome Analysis in Hearing Impaired Patients
Acronym: NGS-NSHL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF96802
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Hearing Impairment
Keywords: Hearing impairment; familial
MeSH Terms: conditions — Hearing Loss | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hearing impaired families: Samples from families presenting with familial hearing impairment, underlying the genetic basis, for whom 74 deafness genes have already been excluded (no evidence of pathogenic genotype)
  Interventions: Genetic: Exome sequencing

INTERVENTIONS:
Genetic: Exome sequencing — DNA extracted from samples will undergo exome sequencing, i.e. sequencing of the coding regions of all known human genes (about 22,000)

SUMMARY:
Hearing impairment is the most frequent sensory deficit in humans and affects one newborn out of 500. The prevalence rises to 3,5/1000 in teenagers due to retarded forms. Most of hearing impairments (about two thirds) have a genetic origin, with recessive, dominant or X-linked mode of inheritance. Some rare forms can be linked to mitochondrial DNA. Molecular diagnosis (i.e. defining the molecular basis of the disease, genes and precise DNA variants) is essential for the follow-up of patients and families.

The project intends to perform exome sequencing on 30 samples of families presenting with hearing impairment. Families have been included based on the genetic origin of the hearing impairment (familial cases) and the exclusion of the involvement of 74 known deafness genes. Exome sequencing (sequencing of the coding regions of all known genes, about 22,000) in these cases may underly new gene/disease relationships.

DETAILED DESCRIPTION:
Exome sequencing will be performed of 10 trios that each include two affected and one non affected members of a family. Filtering of variants will be performed based on frequency. For each trio, data will be analysed in parallel to follow segregation of the variant(s) in candidate genes. The selected candidate genes will be further characterized in order to ascertain their involvement in hearing function.

Finally, once these new genes are well defined as "deafness genes" , their screening will be added to existing diagnostic panels.

ELIGIBILITY:
Inclusion Criteria:

* Families presenting with familial hearing impairment, underlying the genetic basis, for whom 74 deafness genes have already been excluded (no evidence of pathogenic genotype)

Exclusion criteria:

- sporadic cases of hearing impairment, or resolved familial cases

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hearing impaired patients and relatives
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
identification of candidate genes | 1 day
  Description: a candidate gene would present a genotype (combination of DNA variants) compatible with the transmission mode and several lines of evidence of the pathogenic effect of the DNA variants

SECONDARY OUTCOMES:
Quality assessment of the exome sequencing | 1 day
  Quality assessment of the exome sequencing
Quality assessment of the bioinformatics pipelines used | 1 day
  Quality assessment of the bioinformatics pipelines used

CONTACTS AND LOCATIONS:
Overall Officials: Anne Françoise ROUX, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France